CLINICAL TRIAL: NCT07288580
Title: A Phase Ⅰ/Ⅱ, Multicenter, Single-arm, Open-label Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of EHT102 Injection in Pediatric Patients With Biallelic hOTOF Mutations
Brief Title: A Clinical Trial of EHT102 Injection in Pediatric Patients With Biallelic hOTOF Mutations
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Euhearing Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EHT102USCL01; EHT102CNCL02 (Registry Identifier: China)
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Treatment of Congenital Hearing Loss Secondary to Biallelic Mutations of the Otoferlin Gene (OTOF)
Keywords: OTOF

STUDY DESIGN:
Intervention Model Description: EHT102 will be administered as a single intracochlear injection into one or both ears. If bilateral injections are required, they will be performed in a single surgical session
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- The low-dose cohort (Experimental): Participants will receive a single unilateral or bilateral administration of EHT102 at the defined low dose level
  Interventions: Drug: EHT102 Injection
- The high-dose cohort (Experimental): Participants will receive a single unilateral or bilateral administration of EHT102 at the defined high dose level.
  Interventions: Drug: EHT102 Injection

INTERVENTIONS:
Drug: EHT102 Injection — EHT102 injection is a dual-vector gene therapy product developed for the treatment of OTOF-related hearing loss.

SUMMARY:
This study is a multicenter, single-arm, open-label Phase I/II clinical trial, which is designed to evaluate the safety, tolerability and efficacy of EHT102 injection in treating congenital hearing loss secondary to biallelic mutations of OTOF (DFNB9).Up to 30 pediatric participants (A maximum of 15 participants will be enrolled in each of the United States and China) will be enrolled and dosed with EHT102. The dose-escalation phase (Phase I) includes two predefined dose cohorts (3 participants per cohort), with sequential enrollment from low to high dose. During dose escalation, each participant will receive a unilateral EHT102 injection followed by safety observation.

DETAILED DESCRIPTION:
The low-dose and high-dose cohorts will be followed by a 28-day DLT observation period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Prior to study participation, participants and/or their legal guardians must provide informed consent for this trial, voluntarily sign the written informed consent form (ICF), and commit to completing all protocol-specified follow-up visits;
2. Participants must be able to communicate effectively with investigators and comply with study requirements, with guardian assistance if needed. For young children without developed language skills, guardians must ensure cooperation with investigator instructions;
3. Participants and/or their legal guardians must demonstrate adequate comprehension of the trial's nature and maintain realistic expectations regarding potential benefits.
4. Pediatric patients (male or female) aged ≥ 1 and ≤ 17 years at the time of inclusion ;
5. Genetic testing report indicates DFNB9 congenital deafness with Biallelic mutations in the Otoferlin gene;
6. Severe or profound hearing loss (≥65 dB) assessed by ABR, with the sentinel participant having an ABR >90 dB;
7. Meet eligibility criteria for otologic surgery: Absence of middle/inner ear malformations, cochleovestibular nerve abnormalities, or active otologic inflammation as confirmed by computed tomography (CT) and/or magnetic resonance imaging (MRI) within 3 months or during screening period, with surgical suitability determined by the investigator;
8. DPOAE testing shows present response.

Exclusion Criteria:

1. Have other types of hearing loss ineligible for otologic surgery, including but not limited to:

   Middle/inner ear malformations or developmental abnormalities identified by CT/MRI within 3 months; Hearing loss caused by cochleovestibular nerve abnormalities; Conductive hearing loss ; Mixed hearing loss; Syndromic deafness with malformations.
2. Have pre-existing otologic conditions deemed by the investigator to potentially compromise the planned surgery or interfere with study endpoint evaluation, including but not limited to:

   Acute/chronic otitis media;; Ménière's disease; Acoustic neuroma; Unresolved sudden sensorineural hearing loss.
3. Have a history of drug abuse.
4. Have a history of receiving any known ototoxic medications (e.g., aminoglycosides, cisplatin, loop diuretics) within the past 6 months.
5. Antiviral/immunotherapy within 3 months prior to screening.
6. Administration of any live-attenuated vaccines within 30 days prior to screening.
7. Have immunocompromised status or immunodeficiency disorders, including but not limited to:

   Positive HIV antibody (HIV Ab) test; Congenital or acquired immunodeficiency (investigator-determined contraindication to immunosuppressants) ; History of organ transplantation.
8. Have severe systemic diseases or acute conditions, including but not limited to:

   Active tuberculosis; Active herpes zoster infection; Pancreatitis; Renal insufficiency; Gastrointestinal ulcers.
9. Have contraindications to surgery or anesthesia as determined by the surgeon, anesthesiologist, or designated personnel, including but not limited to:

   History of cardiovascular or cerebrovascular events within the past 6 months (e.g., myocardial infarction, heart failure, angina, stroke, or transient ischemic attack) Any other cardiac conditions deemed unsuitable for study participation by the investigator; Known hypersensitivity to the investigational drug.
10. Have participated in gene therapy trials within 6 months prior to screening, plan to participate in other interventional clinical trials within one year post-treatment, or have received investigational drugs within 5 half-lives of the last dose from previous trials.
11. Have implantable devices (e.g., cochlear implants) in the target ear at screening.
12. Have other severe congenital disorders.
13. Have a history of neurological/psychiatric disorders (e.g., epilepsy, dementia).
14. Have chronic anticoagulant therapy that cannot be temporarily discontinued.
15. Have a history of radiotherapy/chemotherapy deemed by investigators to potentially affect trial outcomes.
16. Have tested positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis C virus (HCV) antibody with HCV RNA positive, or positive for human immunodeficiency virus (HIV) antibody, or have active syphilis (TPPA positive and RPR positive).
17. Females of childbearing potential with positive pregnancy tests prior to dosing; Females of childbearing potential and non-sterilized males with fertile partners unwilling/unable to use effective contraception from ICF signing until ≥24 months post-dosing.
18. Any other condition that, at the discretion of the investigator, renders the participant unsuitable for enrollment.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Up to week 52
  Safety will be evaluated by summarizing the number and percentage of participants experiencing treatment-related adverse events (TEAEs) and serious adverse events (SAEs). Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and graded for severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Proportion of Participants Achieving a Hearing Sensitivity Threshold of ≤70 dB by behavioral audiometry | Up to week 26
  This endpoint evaluates the efficacy of EHT102 injection by calculating the percentage of participants who achieve a hearing sensitivity threshold of ≤70 dB in the treated ear, as assessed by behavioral audiometry.

SECONDARY OUTCOMES:
Change from Baseline in Auditory Brainstem Response (ABR) Thresholds | Week 4, Week 13, Week 26, and Week 52
  The change from baseline in ABR thresholds will be assessed in the treated ear. ABR thresholds are measured in decibels (dB). The metric reported will be the change in the average threshold across frequencies (0.5, 1, 2, and 4 kHz) from baseline to each post-treatment time point.
Change from baseline in auditory steady state response (ASSR) thresholds | Week 4, 13, 26, and 52
  This endpoint assesses the change from baseline in Auditory Steady-State Response (ASSR) thresholds in the treated ear. The metric reported will be the mean change in threshold (in dB) across available frequencies from baseline to each post-treatment time point.
Proportion of Participants of a hearing sensitivity threshold of ≤70 dB assessed by behavioral audiometry | Week 4, 13 and 52
  This endpoint evaluates the efficacy of EHT102 injection at additional timepoints by calculating the percentage of participants who achieve a hearing sensitivity threshold of ≤70 dB in the treated ear, as assessed by behavioral audiometry.
Proportion of Participants of a hearing sensitivity threshold of ≤45 dB assessed by behavioral audiometry at Week 26 post injection | Week 26
  This endpoint evaluates a higher efficacy threshold by calculating the percentage of participants who achieve a hearing sensitivity threshold of ≤45 dB in the treated ear at Week 26, as assessed by behavioral audiometry

OTHER OUTCOMES:
Investigator-determined drug/procedure related AEs and SAEs occurring during Years 1-5 post injection | Years 1 through 5
  Long-term safety will be assessed by monitoring the incidence of adverse events (AEs) and serious adverse events (SAEs) that are determined by the investigator to be related to the study drug and/or the surgical procedure during the long-term follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Yilai, M.D. & Ph.D., Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The data generated in this Phase I/II study are proprietary. Aggregate safety and efficacy data will be reported in clinical study reports and potential publications.